CLINICAL TRIAL: NCT05210790
Title: A Phase 3 Study of the Hepcidin Mimetic Rusfertide (PTG-300) in Patients With Polycythemia Vera
Brief Title: A Phase 3 Study of Rusfertide in Patients With Polycythemia Vera
Acronym: VERIFY
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Protagonist Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PTG-300-11
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Polycythemia Vera
Keywords: Polycythemia Vera; PV
MeSH Terms: conditions — Polycythemia Vera

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind (Part 1a):
  Subjects will be randomized in a blinded fashion to 32 weeks of rusfertide or placebo added-on to each subject's ongoing treatment for polycythemia vera.
  Open-label (Part 1b + Part 2):
  Open-label treatment phase during which all subjects who complete Part 1a successfully will receive rusfertide for 124 weeks.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rusfertide (Experimental): Rusfertide (32 Weeks) - Rusfertide (124 Weeks Open-label)
  Interventions: Drug: Rusfertide
- Placebo (Experimental): Placebo (32 Weeks) - Rusfertide (124 Weeks Open-label)
  Interventions: Drug: Placebo; Drug: Rusfertide

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Rusfertide — Experimental drug

SUMMARY:
The study is designed to evaluate the safety and efficacy of rusfertide in subjects with polycythemia vera (PV) in maintaining hematocrit control and in improving symptoms of PV.

DETAILED DESCRIPTION:
Phase 3 study in approximately 250 subjects previously diagnosed with polycythemia vera (PV) who require phlebotomy on a routine basis. There is a 32-week period during which rusfertide or placebo will be added-on to each subject's ongoing therapy for polycythemia vera which may include phlebotomy only or phlebotomy plus stable doses of either of hydroxyurea, interferon and/or ruxolitinib. All subjects who successfully complete the double blind 32-week portion of the study will receive rusfertide for 124 weeks. Approximately 6 and 12 months after their last dose of rusfertide, subjects will have a post-study contact (e.g. by phone) for safety.

ELIGIBILITY:
Main Inclusion Criteria: All subjects must meet ALL of the following inclusion criteria to be enrolled. There are additional inclusion criteria.

* Male and female subjects aged 18 (or the country specific minimum age of consent >18) years or older.
* Meet revised 2016 World Health Organization (WHO) criteria for the diagnosis of polycythemia vera.
* At least 3 phlebotomies due to inadequate hematocrit control in 6 months before randomization or at least 5 phlebotomies due to inadequate hematocrit control in 1 year before randomization.
* CBC values immediately prior to randomization:

  1. Hematocrit <45%,
  2. WBC 4000/μL to 20,000/μL (inclusive), and
  3. Platelets 100,000/μL to 1,000,000/μL (inclusive)
* Subjects receiving cytoreductive therapy at randomization must be on a stable PV therapy regimen.
* Subjects treated with phlebotomy alone at randomization must have stopped cytoreductive therapy 2 to 6 months before screening.

Main Exclusion Criteria: Subjects must meet NONE of the following exclusion criteria to be enrolled. There are additional exclusion criteria.

* Clinically meaningful laboratory abnormalities at Screening.
* Subjects who require phlebotomy at hematocrit levels lower than 45%.
* Clinically significant thrombosis (e.g., deep vein thrombosis or splenic vein thrombosis) within 2 months prior to randomization.
* Active or chronic bleeding within 2 months prior to randomization.
* History of invasive malignancies within the last 5 years, except localized cured prostate cancer and cervical cancer.
* Subjects with in situ or stage 1 squamous cell carcinoma of the skin, in situ or stage 1 basal cell carcinoma of the skin, or in situ melanoma of the skin identified during screen unless the cancer is adequately treated before randomization.
* Received Busulfan, Pipobroman or 32Phosphorus within 7 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving a response who receive rusfertide compared to placebo. | Week 20 through Week 32
  Response is defined as absence of phlebotomy eligibility.

SECONDARY OUTCOMES:
Comparison of mean number of phlebotomies between rusfertide and placebo. | Week 0 to Week 32
Proportion of subjects with HCT values <45% for rusfertide and placebo. | Week 0 to Week 32
Comparison mean change from baseline in total fatigue score based on PROMIS Short Form between rusfertide and placebo. | Week 32
Comparison of mean change from baseline in total MFSAF total score. | Week 32

CONTACTS AND LOCATIONS:
Locations (183):
- United States (79):
  - Infirmary Cancer Care, Mobile, Alabama
  - Palo Verde Hematology-Oncology, Glendale, Arizona
  - City of Hope Medical Center, Duarte, Duarte, California
  - California Cancer Associates for Research and Excellence - Fresno, Fresno, California
  - Marin Cancer Care, Greenbrae, California
  - City of Hope Medical Center, Lenner, Irvine, California
  - University of California, San Diego (UCSD) - Moores Cancer Center, La Jolla, California
  - University of California, Los Angeles (UCLA) - Medical Center, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Sharp Memorial Hospital, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - City of Hope Medical Center, Upland, Upland, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - University of Colorado - Aurora Cancer Center, Aurora, Colorado
  - Rocky Mountain Cancer Centers - Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Rocky Mountain Cancer Centers, Lakewood, Colorado
  - Rocky Mountain Cancer Centers, Littleton, Colorado
  - Rocky Mountain Cancer Centers, Lone Tree, Colorado
  - Yale University School of Medicine - Yale Cancer Center, New Haven, Connecticut
  - BRCR Medical Center, Plantation, Florida
  - BayCare Suncoast Medical Clinic - Hematology/Oncology, St. Petersburg, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Northwest Oncology and Hematology, Rolling Meadows, Illinois
  - Orchard Healthcare Research Inc, Skokie, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Mission Cancer & Blood, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Pontchartrain Cancer Center, Covington, Louisiana
  - Pontchartrain Cancer Center, Hammond, Louisiana
  - American Oncology Partners of Maryland PA (Center for Cancer & Blood Disorders), Bethesda, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Cancer Care Specialists, Reno, Nevada
  - Memorial Sloan Kettering Cancer Center - BASKING RIDGE, Basking Ridge, New Jersey
  - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Memorial Sloan Kettering Cancer Center - MONMOUTH, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center - BERGEN, Montvale, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - New York Cancer and Blood Specialists, Babylon, New York
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center - COMMACK, Commack, New York
  - Memorial Sloan Kettering Cancer Center - WESTCHESTER, Harrison, New York
  - New York Cancer and Blood Specialists, New Hyde Park, New York
  - Memorial Sloan Kettering Cancer Center - KOCH, New York, New York
  - New York Cancer and Blood Specialists, New York, New York
  - Ichan School of Medicine at Mount Sinai, New York, New York
  - New York Presbyterian Hospital/Weill Cornell Medical Center, New York, New York
  - New York Cancer and Blood Specialists, Patchogue, New York
  - New York Cancer and Blood Specialists, Port Jefferson Station, New York
  - New York Cancer and Blood Specialists, Riverhead, New York
  - Wilmot Cancer Institute, University of Rochester, Rochester, New York
  - Montefiore Einstein Center for Cancer Care, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - New York Cancer and Blood Specialists, The Bronx, New York
  - Memorial Sloan Kettering Cancer Center - NASSAU, Uniondale, New York
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - TriHealth Cancer Institute - Good Samaritan Hospital, Cincinnati, Ohio
  - Good Samaritan Infusion Center - Kenwood, Cincinnati, Ohio
  - Good Samaritan Infusion Center - Thomas, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - Oncology Associates of Oregon, Eugene, Oregon
  - Oregon Health and Science University (OHSU) Knight Cancer Institute, Portland, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology San Antonio, San Antonio, Texas
  - Community Cancer Trials of Utah, Ogden, Utah
  - University of Washington - Fred Hutchinson Cancer Center, Seattle, Washington
  - HSHS St. Vincent Hospital, Green Bay, Wisconsin
  - HSHS St. Mary's Hospital, Green Bay, Wisconsin
- Australia (3):
  - One Clinical Research, Nedlands, Perth
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
- Austria (6):
  - Medizinische Universitaet Graz, Graz
  - Kepler Universitaets Klinikum GmbH, Linz
  - Krankenhaus der Elisabethinen Linz, Linz
  - Medizinische Universitaet Wien, Vienna
  - Wiener Gesundheitsverbund-Klinik Hietzing 5-Med., Vienna
  - Klinikum Wels-Grieskirchen Gmb, Wels
- Belgium (3):
  - ZNA Stuivenberg, Antwerp
  - University Hospital Gent, Ghent
  - Campus Gasthuisberg, Leuven
- Canada (4):
  - The University of Alberta - Edmonton, Edmonton, Alberta
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Chile (3):
  - Centro Medico Inmunocel, Las Condes, Santiago Metropolitan
  - Centro de Estudios Clinicos SAGA, Providencia, Santiago Metropolitan
  - Biocenter Centro Clinico de Investigacion, Concepción
- Czechia (3):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Olomouc, Olomouc
  - Vseobecna fakultni nemocnice v Praze, Prague
- France (8):
  - CHU Angers, Angers, Cedex 09
  - AP-HP Hospital Necker-Enfants Malades, Paris, Cedex 15
  - CHU Poitiers, Poitiers, Cedex
  - CHU Amiens Picardie - Hopital Sud, Amiens
  - Centre Hospitalier d'Argenteuil, Argenteuil
  - Centre Hospitalier de Beziers, Béziers
  - AP-HP Hopital Saint-Louis, Paris
  - HCL Centre Hospitalier Lyon Sud, Pierre-Bénite
- Germany (7):
  - Uniklinik RWTH Aachen - Klinik fuer Haematologie, Onkologie, Haemostaseologie und Stammzelltransplantation (Med. Klinik IV), Aachen
  - Charite Universitaetsmedizin Berlin, Berlin
  - Gemeinschaftspraxis Haematologie - Onkologie - Hauptstelle, Dresden
  - Universitaetsmedizin Greifswald, Greifswald
  - ONCOResearch Lerchenfeld GmbH, Hamburg
  - InVo-Institut fuer Versorgungsforschung in der Onkologie GbR, Koblenz
  - Universitaetsmedizin der Johannes Gutenberg - Universitaet Mainz, Mainz
- Queen Mary Hospital, Hong Kong, Hong Kong
- Hungary (3):
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Markhot Ferenc Oktatokorhaz es Rendelointezet, Eger
- Israel (7):
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Center Ein Karem, Jerusalem
  - Shaare Zedek Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center - Davidoff Hematology Center, Petah Tikva
  - Sourasky Medical Center, Tel Aviv
  - Shamir Medical Center (Assaf Harofe), Ẕerifin
- Italy (12):
  - IRCCS Istituto Romagnolo per lo Studio dei Tumori "Dino Amadon", Meldola, Forli-Cesena
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo
  - IRCCS Azienda Ospedaliero-Universtaria di Bologna, Bologna
  - UOC Ematologia - ASST Spedail Civill Brescia, Brescia
  - Azienda Ospedaliero - Universitaria Careggi, Florence
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, SC Ematologia (Padiglione Marcora),, Milan
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - UOC Ematologia e Centro Trapianti AST Pesaro Urbino, Stabilimento Muraglia, Pesaro
  - Fondazione Policlinico Univ. A . Gemelli IRCCS, Roma
  - AOU San Luigi Gonzaga Orbassano, Torino
  - AOU Citta della Salute e della Scienza di Torino, Torino
  - Azienda ASST-SETTELAGHI, Ospedale di Circolo e Fond. Macchi di Varese Ospedael Vecchio, Varese
- Mexico (3):
  - Centro de Estudios de Investigacion SIYODE, Madero
  - SUPERARE Centro de Infusion S.A. de C.V., Mexico City
  - Boca Clinical Trials Mexico S.C. - Ciudad de Mexico, Mexico City
- Netherlands (2):
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Erasmus MC, Rotterdam
- Poland (9):
  - Szpital Specjalistyczny w Brzozowie Podkarpacki Osrodek Onkologiczny im.ks.B.Markiewicza, Brzozów
  - MICS Centrum Medyczne Bydgoszcz, Bydgoszcz
  - Klinika Hematologii I Transplantologii - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Promed P.Lach R.Glowacki Spolka Jawna, Krakow
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Lodzi Oddział, Lodz
  - Wojewodzkie Wielospecjalistyczne Centrum, Onkologii i Traumatologii im. M Kopernika w Lodzi, Lodz
  - MICS Centrum Medyczne Torun, Torun
  - MTZ Clinical Research Powered by Pratia, Warsaw
  - Centrum Medyczne Melita Medical, Wroclaw
- Portugal (4):
  - Conde Hospital Garcia de Orta, Almada
  - Hospital de Braga, Braga
  - CHULN - Hospital de Santa Maria, Lisbon
  - Instituto Portugues de Oncologia do Porto Francisco Gentil, EPE, Porto
- Spain (9):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Hospital Quironsalud de Zaragoza, Zaragoza
- Turkey (Türkiye) (9):
  - Ankara Universitesi Tip Fakultesi Hematologi Bilim dali Ankara, Balkiraz, Ankara
  - Gazi University Medical Faculty, Yenimahalle, Ankara
  - Pamukkale University Hospitals, Pamukkale, Denizli
  - Ege University Hospital Department of Hematology, Bornova, İzmir
  - Karadeniz Technical University Medical Faculty Farabi Hospital, Trabzon, Ortahisar
  - Sanko Universitesi tip Fakultesi Ic Hastaliklari Anabilim Dali, Gaziantep, Sehitkamil
  - Gaziantep Universitesi Sahinbey Arastirma ve Uygulama Hastanesi, Gaziantep
  - Marmara University Pendik Training & Research Hospital, Istanbul
  - Erciyes Universitesi Tip Fakultesi Hastanesi, Dedeman Hospital, Kayseri
- United Kingdom (8):
  - Hillingdon Hospital, Uxbridge, Middlesex
  - Barnet Hospital, Barnet
  - Pilgrim Hospital, Boston
  - Northwick Park Hospital, Harrow
  - The Royal London Hospital, London
  - University College London Hospital, London
  - Royal Free Hospital, Royal Free London NHSFT, London
  - Churchill Hospital, Oxford